CLINICAL TRIAL: NCT03937791
Title: A Phase II Study of Immunotherapy With E7 T Cell Receptor T Cells for Vulvar High-Grade Squamous Intraepithelial Lesions
Brief Title: Immunotherapy With E7 T Cell Receptor T Cells for Vulvar High-Grade Squamous Intraepithelial Lesions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: All analysis with identifiable specimens/data is complete or site has no identifiers linked to the specimens/data. The one enrolled pt has been taken off study
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190091; 19-C-0091
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Squamous Lntraepithelial Lesions of Vulva; Neoplasms, Squamous Cell; Vulvar HSIL
Keywords: Human Papilloma Virus (HPV) Type 16; Retroviral Vector Supernatant; Leukapheresis; T Cell Receptor; Premalignant Epithelial Lesion
MeSH Terms: conditions — Neoplasms, Squamous Cell; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1/1x10^11 E7 T Cell Receptor (TCR) T cells (Experimental): 1x10^11 E7 TCR T cells will be administered intravenously over 20 to 30 minutes on day 0.
  Interventions: Biological: E7 T Cell Receptor (TCR)

INTERVENTIONS:
Biological: E7 T Cell Receptor (TCR) — One dose of E7 TCR T cells (1x10^11 cells) will be administered intravenously over 20 to 30 minutes.

SUMMARY:
Background:

Human papillomavirus (HPV) can cause vulvar high-grade squamous intraepithelial lesions (HSIL). Sometimes, this can become cancer. Researchers want to see if T cell therapy can treat vulvar HSIL. In this therapy, a person s immune cells are genetically modified so they can attack the HPV.

Objective:

To test if a personalized immune treatment can cure vulvar HSIL.

Eligibility:

People ages 18 and older with vulvar HSIL that cannot be removed with surgery, or for which surgery has failed

Design:

Participants will be screened with:

Medical history

Physical exam

HPV testing

Venous assessment

Chest x-ray

Heart and pulmonary tests

Participants will have a baseline visit. They may have a vulvar biopsy. Photographs will be taken of their lesions.

Participants will have leukapheresis: Blood is removed from a needle in the arm and circulated through a machine that takes out the white blood cells. The other blood cells are returned through a needle in the other arm. The white blood cells will be used to grow treatment cells.

Participants will receive the treatment through a tube inserted into an arm, neck, or chest vein. They will recover in the hospital for 1 to 2 days. They will have blood tests and take supportive medications.

Participants may have one more treatment.

Participants will have 5 follow-up visits in the first 3 months after treatment. They may have more visits if their disease is growing. Visits will include blood tests. They may include vulvar biopsies or leukapheresis.

Participants will have an annual physical exam for 5 years after treatment that can be done at home or at the National Institutes of Health (NIH). Then they will have an annual phone or email questionnaire for another 10 years....

DETAILED DESCRIPTION:
Background:

* Vulvar high-grade squamous intraepithelial lesion (HSIL) is a premalignant epithelial lesion that is frequently multifocal and/or recurrent.
* The primary treatment is surgery, which may result in disfigurement and compromise of the urethra, anus, or clitoris. Recurrence after surgery is common and primarily treated with additional surgery.
* Vulvar HSIL is caused by chronic infection with the human papillomavirus (HPV) type 16 infection. In this clinical trial the HPV-16 infection is targeted with a single infusion of autologous T cells that have been genetically engineered to express a HPV-16 E7-specific T cell receptor (E7 TCR T cells).

Objective:

-Determine the complete response rate for E7 TCR T cells in the treatment of vulvar HSIL.

Eligibility:

* Histologically confirmed diagnosis of HPV-16+ vulvar HSIL.
* Expression of the human leukocyte antigen (HLA)-A2*02:01 allele.
* Measurable lesion(s) that are recurrent or cannot be resected with acceptable cosmetic or functional results.
* Age greater than or equal to 18 years old.
* Eastern Oncology Cooperative Group Performance Score of 0 or 1.

Design:

* This is a phase II clinical trial
* Simon minimax two-stage design with initial enrollment of 12 patients and expansion to 16 patients if one or more complete response(s) is/are observed in the initial patients.
* Subjects will receive 1x10^11 E7 TCR T cells
* No conditioning regimen or aldesleukin will be given
* Re-enrollment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have vulvar High-Grade Squamous Intraepithelial Lesions (HSIL) as confirmed by pathology report from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
* Vulvar HSIL must be human papillomavirus (HPV)-16+ by a polymerase chain reaction (PCR), Ribonucleic acid (RNA), or in situ hybridization test from a CLIA certified laboratory.
* Patients must have measurable lesion(s) as defined in one or more of the following criteria:

  * Failure of surgery to control disease (i.e. positive margins after surgery or recurrence of HSIL after surgery).
  * Multifocal or extensive disease for which surgery would result in disfigurement that is not be acceptable to the patient.
  * Disease for which surgery would have a risk of functional impairment that is not be acceptable to the patient (i.e. involve partial or complete excision of the clitoris, anus, vagina, or urethra).
* Patients may have received any previous therapy, including surgical excision. Patients with recurrent disease must have histologically documented recurrence on new biopsy and a measurable lesion that meets the above criteria.
* Patients must have the human leukocyte antigen (HLA)-A*02:01 allele
* Age greater than or equal to18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Able to understand and sign the Informed Consent Document.
* Women of child-bearing potential must have a negative pregnancy test. Women of child-bearing potential are defined as all women who are not post-menopausal or who have not had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* The effects of E7 T-Cell Receptor (TCR) T Cells on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Seronegative for human immunodeficiency virus (HIV) antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment.
* Seronegative for hepatitis B antigen and hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by reverse transcription (RT)-PCR and be hepatitis C virus (HCV) RNA negative.
* Must be willing to participate in Gene Therapy Long Term Followup Protocol (20-C-0051), which will follow patients for up to 15 years per Food and Drug Administration (FDA) requirements.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin greater than or equal to 9.0 g/dL
  * total bilirubin within 1.5X normal institutional limits except in patients with Gilbert's Syndrome who must have a total bilirubin < 3.0 mg/dL
  * Aspartate Aminotransferase (AST)/Serum glutamic-oxaloacetic transaminase(SGOT)/Alanine Aminotransferase (ALT)/Serum glutamic pyruvic transaminase,(SGPT) Serum ALT/AST < 3X upper limit of normal (ULN)
  * creatinine < 1.5X baseline, < 1.5X ULN OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR, breastfeeding should be discontinued if the mother is treated with E7 TCR. These potential risks may also apply to other agents used in this study.
* Uncontrolled intercurrent illness including, but not limited to, any ongoing or active infection (e.g. requiring anti-infective therapy), coagulation disorders, cardiovascular disorders, respiratory disorders, cancer, or psychiatric illness/social situations (within the last six months) that would limit compliance with study requirements.
* Any form of systemic immunodeficiency, including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence maybe less responsive to the treatment.
* Concurrent systemic steroid therapy if greater than the equivalent of 5 mg prednisone by mouth (PO) daily. Patients previously on steroids must be off steroids for four weeks prior to treatment.
* Cardiac stress test and pulmonary function tests maybe required for patients with a clinical history of significat cardiopulmonary disease. Patients with active cardiac ischemia or severe chronic obstructive pulmonary disease are not eligible.
* Patients with any active invasive cancer are not eligible.
* Patients with vulvar HSIL that is not HPV-16+ or is associated with multiple types of high-risk HPV at the time of eligibility assessment are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0091.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Participants With Vulvar High-Grade Squamous Intraepithelial Lesions (HSIL) Who Experience a Complete Response for E7 T-Cell Receptor (TCR) T Cells Treatment
Description: The fraction of patients who experience a complete response. Complete Response is disappearance of all target lesions. No appearance of new lesions.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 1
Proportion of participants | 0

2. Secondary Outcome: Number of Grade 2 Adverse Events Unlikely Related to Drug in Participants Who Received E7 T-Cell Receptor (TCR) T Cells Administered in a Low Intensity Setting Without Conditioning or Systemic Aldesleukin
Description: Grade 2 adverse event is moderate.
Time Frame: 30 days following the last dose of study therapy
Measure: Number; unit: adverse events
Arm/Group | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 1
adverse events | 1

3. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 6 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 6 days.
Arm/Group | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/1x10^11 E7 T Cell Receptor (TCR) T Cells (N=1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03937791/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort Screening Consent (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT03937791/ICF_001.pdf
  • Informed Consent Form: Cohort Treatment Consent (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT03937791/ICF_002.pdf